CLINICAL TRIAL: NCT07066293
Title: Evaluation of Using Sticky Bone Grafting Combined With Concentrated Growth Factor Membrane for Repair of Unilateral Alveolar Cleft
Brief Title: Sticky Bone Grafting With Concentrated Growth Factor Membrane for Repair of Unilateral Alveolar Cleft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Maram Nashaat Breshah, Lecturer of Oral & Maxillofacial Surgery, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #R-OS-11-22-2
Record Dates: First submitted 2025-07-04; First posted 2025-07-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-07

CONDITIONS: Unilateral Alveolar Cleft of Maxilla
Keywords: alveolar cleft; sticky bone; concentrated growth factor; volumetric assessment; bone mineral density

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sticky Bone grafting with concentrated growth factor membrane for unilateral alveolar cleft (Experimental): This will include 10 patients in whom unilateral alveolar cleft will be repaired using sticky bone grafting combined with concentrated growth factor membrane
  Interventions: Procedure: Unilateral alveolar cleft repair

INTERVENTIONS:
Procedure: Unilateral alveolar cleft repair — 10 patients in whom unilateral alveolar cleft will be repaired using sticky bone grafting combined with concentrated growth factor membrane

SUMMARY:
The aim of this study is to evaluate using Sticky Bone grafting combined with concentrated growth factor membrane for repair of unilateral alveolar cleft.

DETAILED DESCRIPTION:
This study will be carried out on ten patients with unilateral alveolar clefts, The patients will be recieved, clinically& radiographically examined and managed at Oral & Maxillofacial Surgery Department, Faculty of Dentistry, Tanta University.

Preoperative evaluation:

Clinical evaluation will include presence of oronasal fistulas, nasal regurgitation and Presence of erupting teeth in cleft. .Preoperative cone beam computed tomography (CBCT) scans will be analyzed to measure alveolar cleft dimensions and the total cleft defect volume will be calculated.

Surgical technique:

Under general anesthesia, mucoperiosteal flaps will be raised along the cleft margins, exposing the defect. The nasal lining will be sutured with 4/0 Vicryl, followed by the application of a concentrated growth factor (CGF) membrane to cover the nasal mucosa. The sticky bone graft will be packed tightly into the cleft, ensuring complete defect filling. A CGF membrane will be then placed over the graft to enhance stability and healing. The flaps will be sutured using tension-free interrupted 3/0 Vicryl sutures to ensure full coverage of the graft.

Postoperative evaluation:

The patients will be evaluated over a nine-months follow-up period clinically at intervals of 1st & 2nd weeks, then 1st ,3rd and 9th months for healing parameters such as infection, wound dehiscence, recurrence of oronasal fistulas, nasal regurgitation and graft exposure & radiographically by using CBCT for assessing graft volume, bone mineral density immediate, 3rd & 9th months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral alveolar clefts requiring repair.
* patients free from any systemic disease that may affect normal healing of bone.
* patients at an age older than 12 years

Exclusion Criteria:

* Bilateral alveolar clefts.
* Immunocompromised patients.
* Syndromic patients.

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-10-02 (Actual)

PRIMARY OUTCOMES:
inflammation | 1 month
  mild, moderate, severe
nasal regurgitation | 1 month
  Yes or No
fistula recurrence | 1 month
  positive or negative
bone graft volume | 1 month
  soft ware
bone mineral density | 1 month
  soft ware

SECONDARY OUTCOMES:
bone graft volume | 9 months
  soft ware
bone mineral density | 9 months
  soft ware

CONTACTS AND LOCATIONS:
Overall Officials: Omnia M Saber, Principal Investigator — Faculty of Dentistry, Tanta University, Egypt; Mohamed S Khedr, Prof, Principal Investigator — Faculty of Dentistry, Tanta University, Egypt; Ahmed M Elshareef, Ass prof, Principal Investigator — Faculty of Dentistry, Tanta University, Egypt; Maram N Breshah, Lecturer, Principal Investigator — Faculty of Dentistry, Tanta University, Egypt
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No